CLINICAL TRIAL: NCT01522599
Title: Flow-flow ECCO2-R and 4 ml/kg Tidal Volume vs. 6 ml/kg Tidal Volume to Enhance Protection From Ventilator Induced Lung Injury in Acute Lung Injury (ELP)
Brief Title: Flow-flow ECCO2-R and 4 ml/kg Tidal Volume vs. 6 ml/kg Tidal Volume to Enhance Protection From VILI in Acute Lung Injury
Acronym: ELP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Financial hardship
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Marco Ranieri, Principal Investigator, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELP-CEI315
Record Dates: First submitted 2012-01-26; First posted 2012-01-31 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS: Acute Respiratory Distress Syndrome; LOW FLOW ECCO2-R: EXTRA-CORPOREAL CO2 REMOVAL; VILI: Ventilator Induced Lung Injury
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARDS-Net strategy (Control) (Active Comparator)
  Interventions: Other: ARDS-Net Strategy
- ECCO2-R with 4 mL/Kg Vt (Treatment) (Experimental)
  Interventions: Other: ECCO2-R

INTERVENTIONS:
Other: ARDS-Net Strategy — Treatment according to the ARDS-Net protocol (The Acute Respiratory Distress Syndrome Network N Engl J Med 2000; 342:1301-1308May 4, 2000)
  Other Names: Protective ventilation
  Arms: ARDS-Net strategy (Control)
Other: ECCO2-R — Ventilation with Tidal Volume of 4 ml/kg PBW and low flow CO2 removal
  Other Names: Further protective ventilation
  Arms: ECCO2-R with 4 mL/Kg Vt (Treatment)

SUMMARY:
The main objective of this randomized multicenter clinical trial is to test the hypothesis that further reduction of VT to 4mL/kg may enhance lung protection in patients with ARDS as compared to the conventional "ARDS-Net" ventilation. Control of PaCO2 in the ~4 ml/kg arm would be accomplished by LFPPV- ECCO2-R.

DETAILED DESCRIPTION:
The trial will test the hypothesis that a VT of 4 ml/kg PBW combined with low flow CO2 removal improves outcome in patients with severe ARDS (PFs ≤ 200 and PEEP ≥ 10) compared to ventilation with a VT of 6 ml/kg PBW. The study will accrue a maximum of 230 patients over approximately 12-18 months.

PRIMARY END-POINT: Number of ventilator-free days (VFDs) during the 28 days immediately after randomization

SECONDARY END-POINTS: 28 and 90-day all-cause mortality; number of ICU-free days during the 28 days immediately after randomization; cumulative incidence of: first episode of refractory hypoxemia (during 28 days after randomization), use of rescue therapies, first day that meet criteria for weaning, SOFA-free and severe adverse events.

Patients in CONTROL will be treated according to a modified, simplified version of The ARDS-Network lung protective lower tidal volume. Patients in TREATMENT group will be treated according to the ARDS-Net protocol modified (VT reduced by 1 ml/kg PBW at intervals ≤ 2 hours until VT = 4ml/kg PBW and the use of low-flow CO2 removal with a Plateau Pressure Goal: ≤ 25 cm H2O).

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* are on invasive assisted breathing less then 48 hours
* less than 24 hours since diagnosis for ARDS: with PF<=200 and PEEP>=10, bilateral infiltrate on chest X-Ray and no clinical evidence of left atrial hypertension
* have a commitment to full support

Exclusion Criteria:

* intubation and mechanical ventilation (any form) for > 48 hours
* risk of systemic bleeding with anticoagulation
* acute brain injury
* body mass index > 40
* neuromuscular disease that impairs ability to ventilate without assistance
* severe chronic respiratory disease
* burns > 40% total body surface area
* malignancy or other irreversible disease or condition for which 6- month mortality is estimated to be greater than 50%
* allogeneic bone marrow transplant within the last 5 years
* chronic respiratory condition making patient respirator dependent
* patient, surrogate, or physician not committed to full support
* acute myocardial infarction or acute coronary syndrome within 30 days
* moribund patient: not expected to survive 24 hours
* no consent/inability to obtain consent
* patients receiving high frequency ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2012-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Number of ventilator-free days during the 28 days immediately after randomization | 28 DAYS
  VFDs is a composite endpoint. VFD to day 28 is defined as the number of days after initiating unassisted breathing to day 28 after randomization, assuming a patient survives for at least two consecutive calendar days after initiating nassisted breathing and remains free of assisted breathing. If a patient dies prior to day 28 or is still receiving assisted breathing at day 27, his/her VFDs will be zero.

SECONDARY OUTCOMES:
28-day all-cause mortality | 28 days
  All patients will be classified as either "alive at Study Day 28" or, if dead, "dead at Study Day 28." For example, day zero is the day of randomization and day 1 is the next day and encompasses all events that occur midnight-to-midnight, etc.
90-day all-cause mortality. | 90 days
  All patients will be classified as either "alive at Study Day 90" or, if dead, "dead at Study Day 90. Patients alive in hospital or in any health care facility at day 90 will be considered to have survived.
Number of ICU-free days during the 28 days immediately after randomization (ICU-FD). | 28 days
  ICU-FDs are defined as the number of days from the time of ICU discharge to day 28 after randomization, assuming survival for at least two consecutive calendar days after ICU discharge and continued stay outside the ICU setting to day 28. If a patient returns to the ICU and subsequently needs ICU admission to day 28, ICU-FDs will be counted from the end of the last period of ICU discharge to day 28.
Cumulative incidence of first episode of refractory hypoxemia (during 28 days after randomization). | 28 days
  Refractory hypoxemia is defined as PaO2 < 60 mm Hg for at least 1 hour while receiving an FIO2 of 1.0
Cumulative incidence of the use of rescue therapies. | 28 days
  The first day inhaled nitric oxide or prone position or high-frequency oscillation or high-frequency oscillatory ventilation or extracorporeal membrane oxygenation or any combinations of these therapies will be tabulated.
Cumulative incidence of first day that meet criteria for weaning readiness during 28 days after randomization. | 28 days
  Weaning readiness will be defined if the following 4 criteria are met for the last 30 minutes during a spontaneous breathing trial (SBT).
  1. SpO2 ≥ 90% and / or PaO2 ≥ 60 mm Hg; PaO2 to take precedence if both available
  2. Respiratory Rate ≤ 35 / min
  3. pH ≥ 7.30
  4. No respiratory distress
Cumulative SOFA-free score between randomization and day 28. | 28 days
  The SOFA-free score is calculated as the maximum daily score, minus the observed SOFA score. To monitor the degree of variation of the patient's SOFA score (as improvement or worsening) the daily difference between the maximum score and the observed score will be summed up for each day between randomization and day 28. Patients dying before the 28th day cannot continue to increase their cumulative SOFA-free score. In this way, the larger the cumulative score reached, the higher is the improvement of the patient and the probability of being alive at day 28.
Cumulative incidence of severe adverse events during 28 days after randomization. | 28 days
  Adverse events that are considered to be related to ECCO2-R and that follows a reasonable temporal sequence from the ECCO2-R and that could readily have been produced by ECCO2-R will be classified as: "DEVICE RELATED" or "PATIENT RELATED"

CONTACTS AND LOCATIONS:
Overall Officials: Vito Marco VM Ranieri, MD, Principal Investigator — Department of Anesthesia and Intensive Care Medicine, University of Turin, Italy; Antonio A Pesenti, MD, Study Chair — Department of Perioperative Medicine and Intensive Care, San Gerardo Hospital, Monza, Italy
Locations (1):
- University of Turin - Department of Anesthesia and Intensive Care Medicine, Turin, Italy